CLINICAL TRIAL: NCT00598234
Title: Perioperative Pain Control With Celecoxib (Celebrex) in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ching-Chuan Jiang, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 950704
Record Dates: First submitted 2008-01-10; First posted 2008-01-21 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Celecoxib (Celebrex)
  Interventions: Drug: Celecoxib (Celebrex)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Celecoxib (Celebrex)

INTERVENTIONS:
Drug: Celecoxib (Celebrex) — The study group received 400mg oral celecoxib about 1 hr prior to surgery, and 200mg every 12 hrs, along with PCA morphine, over the first five post-operative days. The control group received placebo, along with PCA morphine over the same postoperative period. All patients received Acetaminophen 500mg qid for pain control.

SUMMARY:
We propose that administration perioperative celecoxib is effective to control postoperative VAS pain scores, improve rehabilitation results, and decrease narcotics usage in total knee replacement patients.

DETAILED DESCRIPTION:
Total knee replacement is an effective method to treat end-stage osteoarthritis. However, post-operative pain is still a bothering problem. Pre-emptive analgesia is defined as an antinociceptive treatment which prevents pain before its onset. Preoperative analgesia is thought more effective than an equal post-operative dose. Surgical trauma induces the synthesis of prostaglandins, which sensitize the peripheral nociceptors.Non-steroidal anti-inflammatory drugs (NSAIDs) inhibit prostaglandin synthesis both in the periphery and the spinal cord, therefore decreasing the post-operative hyperalgesic state.

Celebrex (Celecoxib) is a nonsteroidal anti-inflammatory drug (NSAID) that is used to treat arthritis, pain, menstrual cramps, and colonic polyps. Prostaglandins are chemicals that are important contributors to the inflammation of arthritis that causes the pain, fever, swelling and tenderness. Celecoxib blocks the enzyme that makes prostaglandins (cyclooxygenase 2), resulting in lower concentrations of prostaglandins. As a consequence, inflammation and its accompanying pain, fever, swelling and tenderness are reduced. Celecoxib differs from other NSAIDs in that it causes less inflammation and ulceration of the stomach and intestine (at least with short-term treatment) and does not interfere with the clotting of blood.

The study group received 400mg oral celecoxib about 1 hr prior to total knee replacement surgery, and 200mg every 12 hrs, along with PCA morphine, over the first five post-operative days. The control group received placebo, along with PCA morphine over the same postoperative period. All patients had spinal anesthesia and hemovac drain tubes inserted for postoperative blood loss evaluation.

Specific aims and goals:

1. to establish better rehabilitation results and lower VAS pain scores after administration perioperative celecoxib in total knee replacement patients.
2. to establish morphine sparing effect after perioperative celecoxib administration.
3. to evaluate the risks after prescribing perioperative celecoxib.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving total knee replacement will be recruited in this study.

Exclusion Criteria:

* subjects with end-stage renal disease, cerebral vascular accident, peptic ulcer, long-term usage of NSAIDs.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
VAS pain scores, range-of-motion, narcotics usage | post-op 6hrs,12hrs,day1,day2,day3,day7

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Chuan Jiang, M.D.;Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- Ching-Chuan Jiang, Taipei, Taiwan

REFERENCES:
- [Derived] Huang YM, Wang CM, Wang CT, Lin WP, Horng LC, Jiang CC. Perioperative celecoxib administration for pain management after total knee arthroplasty - a randomized, controlled study. BMC Musculoskelet Disord. 2008 Jun 3;9:77. doi: 10.1186/1471-2474-9-77. PMID 18519002